CLINICAL TRIAL: NCT03669380
Title: Isolated Superior Mesenteric Artery Dissection With Concomitant Vascular Aberrancy: Extremely Rare Cases and Clinical Implications
Brief Title: Superior Mesenteric Artery Dissection
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Lei Dou, principal investigator, Tongji Hospital
Other Study IDs: TJ-207101
Record Dates: First submitted 2018-05-12; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- conservative treatment: Conservative treatment consisted of bowel rest, intravenous fluid therapy, nutritional support, strict blood pressure control, anticoagulation (with or without antiplatelet) and close observation
- Interventional and surgical treatment: Interventional and surgical treatment

INTERVENTIONS:
Other:
  Groups: Interventional and surgical treatment

SUMMARY:
This study investigate CT images of patients with spontaneous isolated superior mesenteric artery dissection (SISMAD). The investigators also further analyze the CT morphological differences between different options, aiming to determine "alarming CT character" during initial conservative treatment.

DETAILED DESCRIPTION:
57 Patients with SISMAD from Oct 2011 to Jan 2018 in investigator's hospital were included in this research. The investigators collected relevant clinical data and further investigated the CTA characters of both true lumen and false lumen. SMA angle, distance between entry site of dissection and SMA root were also measured.

ELIGIBILITY:
Inclusion Criteria:

* SMA dissection

Exclusion Criteria:

* SMA dissection combined with aortic or other visceral arteries
* Trauma related SMA dissection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between Oct. 2011 and Jan. 2018, a total of 57 consecutive patients with SISMAD were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Diameters of true lumen | up to 6 months
  Measure the diameters of patent true lumen in patients with isolated mesenteric artery dissection
  thrombosis in the false lumen , the distance between entry site of dissection and SMA root (P=0.133), the presence of SMA branch involving (P=0.322) have no difference in different treatment groups
the distance between dissection and SMA root | up to 6 months
  Measure the distance between dissection and SMA root in patients with isolated mesenteric artery dissection
the angle between SMA root and abodominal aorta | up to 6 months
  Measure the angle between SMA root and abodominal aorta in patients with isolated mesenteric artery dissection

CONTACTS AND LOCATIONS:
Overall Officials: Lei Dou, Dr., Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No